CLINICAL TRIAL: NCT03976921
Title: Impact of Stress Cardiac Computed Tomography Myocardial Perfusion on Downstream Resources and PROgnosis in Patients With Suspected or Known Coronary Artery Disease: a Multicenter International Study
Brief Title: Impact of Stress CT Myocardial Perfusion on Downstream Resources and Prognosis
Acronym: CTP-PRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Medical University of South Carolina (Other); Semmelweis University Heart and Vascular Center (Other); Emory University (Other); UMC Utrecht (Other); Johns Hopkins University (Other); Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Pontone, MD, PhD, Director of MR Unit & Deputy Director of Cardiovascular CT Unit, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R993/19-CCM 1044
Record Dates: First submitted 2019-05-30; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Computed Tomography Perfusion; Cardiovascular Outcomes; Cost-effectiveness
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Upon completion of the screening procedure and enrollment, the patients will be randomized 1:1 to the CT-based strategy (Group A) or usual care (Group B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCTA Strategy (Experimental): CCTA will be performed with one of the latest generation scanners. A stenosis > 50% will be considered as significant from an anatomical point of view. For coronary stents, degree of intrastent restenosis will be evaluated by visual assessment of intraluminal contrast density. ISR > 50% will be considered as significant from an anatomical point of view. For CABG, each graft will be visually evaluated and scored as patent, non-significant stenosis ≤ 50%, significant stenosis > 50%, or occluded. For patients with positive CCTA results, additional stress CTP will be performed subsequently. If indicated, vasodilatation will be induced with i.v. adenosine injection or regadenoson. Static or dynamic CTP will be performed according to local practice and scanner technology available. For all patients with previous history of MI the presence of reversible ischemia will be obtained by the comparison between rest and stress perfusion.
  Interventions: Diagnostic Test: Integration of CCTA with stress CTP when indicated
- Standard of care Strategy (Active Comparator): Patients randomized to this group will be evaluated according to current clinical guidelines with the following approaches: (a) stress ECG, or imaging-based tests such as Stress Echo, Stress CMR, SPECT or PET; (b) direct referral to ICA.
  Interventions: Diagnostic Test: Standard of care approach

INTERVENTIONS:
Diagnostic Test: Integration of CCTA with stress CTP when indicated — When judged indicated, functional assessment with stress CTP perfusion will be performed on top of CCTA.
  Arms: CCTA Strategy
Diagnostic Test: Standard of care approach — (a) functional non-invasive tests (stress ECG, or imaging-based tests such as Stress Echo, Stress CMR, SPECT or PET) as a gatekeeper for ICA; (b) direct referral to ICA.
  Arms: Standard of care Strategy

SUMMARY:
CT myocardial perfusion imaging (CTP) represents one of the newly developed CT-based techniques but its cost-effectiveness in the clinical pathway is undefined. The aim of the study is to evaluate the usefulness of combined evaluation of coronary anatomy and myocardial perfusion in intermediate to high-risk patients for suspected CAD or with known disease in terms of clinical decision-making, resource utilization and outcomes in a broad variety of geographic areas and patient subgroups.

DETAILED DESCRIPTION:
The use of cardiac computed tomography angiography (CCTA) is usually suggested in low to intermediate risk for its diagnostic and prognostic role to rule out CAD with low radiation exposure. In the setting of intermediate to high risk patients, the addition of functional information is prognostically useful and, in patients with previous history of percutaneous coronary intervention (PCI), functional strategy has been shown to be more cost-effective as compared to anatomical assessment CT myocardial perfusion imaging (CTP) represents one of the newly developed CT-based techniques, combining both anatomical and functional evaluation of CAD in a single imaging modality. More recently, stress CTP was shown to provide additional diagnostic value as compared to CCTA alone in intermediate to high risk patients. The purpose of this study will be to evaluate the usefulness and impact of combined evaluation of coronary artery anatomy and myocardial perfusion with CCTA+CTP in intermediate to high risk patients for suspected CAD or with known disease in terms of clinical decision-making, resource utilization, and outcomes in a broad variety of geographic areas and patient subgroups.

CTP-PRO study is a cooperative, international, multicentre, prospective, open-label, randomized controlled study evaluating the cost-effectiveness of a CCTA+CTP strategy versus usual care in intermediate to high risk patients with suspected or known CAD who undergo clinically indicated diagnostic evaluation.

Patients will be screened for study eligibility. Patients meeting all selection criteria will be asked to sign an informed consent document prior to undergoing any study-specific evaluation; then a structured interview will be performed and a clinical history obtained, assessing the presence of common cardiac risk factors, drug therapy (focus on statin, aspirin and/or antiplatelet agent use) and symptoms (typical or atypical angina, to estimate the pre-test likelihood of CAD).

Upon completion of the screening procedure and enrollment, the patients will be randomized 1:1 to the CT-based strategy (Group A) or usual care (Group B). Patient follow-up will be performed at 1 year (± 1 month) and 2 years (± 1 month) by trained interviewers who check medical records or by phone interview collecting the following information: downstream testing; overall radiation exposure; outcomes; cost-effectiveness estimation.

The primary endpoint of the study is the reclassification rate of CCTA in group B due to the addition of CTP. The secondary endpoint will be the comparison between group A and group B in terms of non-invasive and invasive downstream testing, prevalence of obstructive CAD at ICA, revascularization, cumulative ED and overall cost during the follow-up at 1- and 2-years. The tertiary endpoint will be the comparison between each group in terms of MACE and cost-effectiveness at 1- and 2-years.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (age ≥ 18 years) with known or suspected CAD referred for clinically indicated diagnostic evaluation.
* CCTA has to be performed with the state of art in terms of scanner technology as follow: Revolution CT (GE Healthcare, Milwaukee, WI), CardioGraphe (Arineta, Caesarea, Israel), SOMATOM Force (Siemens, Forchheim, Germany), Brilliance iCT and IQon CT (Philips, Best, Netherlands), Aquilion One Vision (Toshiba Medical Systems Corp., Otawara, Japan).

Exclusion Criteria:

* Performance of any non-invasive diagnostic testing within 90 days before enrollment
* Low to intermediate pre-test likelihood of CAD according to the updated Diamond-Forrester risk model score
* Acute coronary syndrome
* Need for an emergent procedure
* Evidence of clinical instability
* Contra-indication to contrast agent administration and/or impaired renal function
* Inability to sustain a breath hold
* Pregnancy
* Cardiac arrhythmias
* Presence of pace maker or implantable cardioverter defibrillator
* Contra-indications to the administration of sub-lingual nitrates, beta-blockade and adenosine
* Structural cardiomyopathy outside of suspected or know ischemic heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Reclassification rate of CCTA in group B due to the addition of CTP | 30 days.
  For each enrolled patient in whom both CCTA and stress CTP will be performed, the endpoint review committee will use data from coronary CTA and CTP, along with the clinical data to determine the management plan using the following criteria: (a) optimal medical therapy, (b) more non-invasive information required, (c) invasive evaluation required, (d) revascularization treatment (PCI or CABG or hybrid treatment).

SECONDARY OUTCOMES:
Downstream non-invasive testing | 1- and 2-years.
  Comparison between group A and group B in terms of number of non-invasive downstream testing (Exercise EKG, Stress-Echo, SPECT, Stress CMR, PET) or invasive testing (invasive coronary angiography) performed after the randomization.
Downstream invasive testing | 1- and 2-years.
  Comparison between group A and group B in terms of number of downstream invasive testing (invasive coronary angiography) performed after the randomization.
Prevalence of obstructive CAD at ICA | 1- and 2-years.
  Comparison between group A and group B in terms of number of patients with obstructive CAD at ICA.
Revascularization | 1- and 2-years.
  Comparison between group A and group B in terms of number of patients treated with revascularization (PCI or CABG or hybrid treatment).
Effective Dose | 1- and 2-years.
  Comparison between group A and group B in terms of cumulative Effective Dose (ED), measured in mSv, due to non-invasive or invasive testing performed after randomization.
Overall costs related to downstream diagnostic tests. | 1- and 2-years.
  Comparison between group A and group B in terms of overall costs of downstream diagnostic tests (sum of costs of all diagnostic tests performed after randomization), expressed in Dollars, according to local reimbursement.

OTHER OUTCOMES:
Hospitalization for cardiac reason | 1- and 2-years.
  Comparison between group A and group B group in terms of number of patients that needed hospitalization for cardiac reason.
Unstable angina | 1- and 2-years.
  Comparison between group A and group B group in terms of number of patients that needed hospitalization for unstable angina (defined according to 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J 2016:37,267-315).
Non-fatal myocardial infarction | 1- and 2-years.
  Comparison between group A and group B group in terms of number of patients that experienced non-fatal myocardial infarction (defined according to Fourth universal definition of myocardial infarction, 2018. Eur Heart J 2019:40,237-269).
Cardiac death | 1- and 2-years.
  Comparison between group A and group B group in terms of number of patients that experienced death because of immediate cardiac cause (e.g., MI, low-output failure, fatal arrhythmia) or vascular cause (e.g., cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause). Unwitnessed death and death of unknown cause will be classified as cardiovascular death.
MACE (Major adverse cardiovascular events) | 1- and 2-years.
  MACE will be defined as a combined endpoint of unstable angina, nonfatal MI, and cardiac death.
Cost-effectiveness ratio | 1- and 2-years.
  Cost-effectiveness ratio will be calculated according to the following equation: (Index test cost + downstream diagnostic tests cost) / projected remaining life expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Pontone, MD, PhD, Principal Investigator — Centro Cardiologico Monzino, IRCCS; U. Joseph Schoepf, MD, Principal Investigator — Medical University of South Carolina

REFERENCES:
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Pijls NH, Fearon WF, Tonino PA, Siebert U, Ikeno F, Bornschein B, van't Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, De Bruyne B; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention in patients with multivessel coronary artery disease: 2-year follow-up of the FAME (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation) study. J Am Coll Cardiol. 2010 Jul 13;56(3):177-84. doi: 10.1016/j.jacc.2010.04.012. Epub 2010 May 28. PMID 20537493
- [Background] Shaw LJ, Berman DS, Maron DJ, Mancini GB, Hayes SW, Hartigan PM, Weintraub WS, O'Rourke RA, Dada M, Spertus JA, Chaitman BR, Friedman J, Slomka P, Heller GV, Germano G, Gosselin G, Berger P, Kostuk WJ, Schwartz RG, Knudtson M, Veledar E, Bates ER, McCallister B, Teo KK, Boden WE; COURAGE Investigators. Optimal medical therapy with or without percutaneous coronary intervention to reduce ischemic burden: results from the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial nuclear substudy. Circulation. 2008 Mar 11;117(10):1283-91. doi: 10.1161/CIRCULATIONAHA.107.743963. Epub 2008 Feb 11. PMID 18268144
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Pontone G, Muscogiuri G, Baggiano A, Andreini D, Guaricci AI, Guglielmo M, Fazzari F, Mushtaq S, Conte E, Annoni A, Formenti A, Mancini E, Verdecchia M, Fusini L, Bonfanti L, Consiglio E, Rabbat MG, Bartorelli AL, Pepi M. Image Quality, Overall Evaluability, and Effective Radiation Dose of Coronary Computed Tomography Angiography With Prospective Electrocardiographic Triggering Plus Intracycle Motion Correction Algorithm in Patients With a Heart Rate Over 65 Beats Per Minute. J Thorac Imaging. 2018 Jul;33(4):225-231. doi: 10.1097/RTI.0000000000000320. PMID 29346192
- [Background] Erthal F, Premaratne M, Yam Y, Chen L, Lamba J, Keenan M, Haddad T, Pharasi K, Anand S, Beanlands RS, Burwash IG, Dwivedi G, Ruddy TD, Chow BJW. Appropriate Use Criteria for Cardiac Computed Tomography: Does Computed Tomography Have Incremental Value in All Appropriate Use Criteria Categories? J Thorac Imaging. 2018 Mar;33(2):132-137. doi: 10.1097/RTI.0000000000000297. PMID 28914747
- [Background] Pontone G, Bertella E, Mushtaq S, Loguercio M, Cortinovis S, Baggiano A, Conte E, Annoni A, Formenti A, Beltrama V, Guaricci AI, Andreini D. Coronary artery disease: diagnostic accuracy of CT coronary angiography--a comparison of high and standard spatial resolution scanning. Radiology. 2014 Jun;271(3):688-94. doi: 10.1148/radiol.13130909. Epub 2014 Feb 8. PMID 24520943
- [Background] Pontone G, Andreini D, Bartorelli AL, Bertella E, Cortinovis S, Mushtaq S, Foti C, Annoni A, Formenti A, Baggiano A, Conte E, Bovis F, Veglia F, Ballerini G, Fiorentini C, Agostoni P, Pepi M. A long-term prognostic value of CT angiography and exercise ECG in patients with suspected CAD. JACC Cardiovasc Imaging. 2013 Jun;6(6):641-50. doi: 10.1016/j.jcmg.2013.01.015. PMID 23764093
- [Background] Pontone G, Andreini D, Guaricci AI, Rota C, Guglielmo M, Mushtaq S, Baggiano A, Beltrama V, Fusini L, Solbiati A, Segurini C, Conte E, Gripari P, Annoni A, Formenti A, Petulla' M, Lombardi F, Muscogiuri G, Bartorelli AL, Pepi M. The STRATEGY Study (Stress Cardiac Magnetic Resonance Versus Computed Tomography Coronary Angiography for the Management of Symptomatic Revascularized Patients): Resources and Outcomes Impact. Circ Cardiovasc Imaging. 2016 Oct;9(10):e005171. doi: 10.1161/CIRCIMAGING.116.005171. PMID 27894070
- [Background] Schuijf JD, Wijns W, Jukema JW, Atsma DE, de Roos A, Lamb HJ, Stokkel MP, Dibbets-Schneider P, Decramer I, De Bondt P, van der Wall EE, Vanhoenacker PK, Bax JJ. Relationship between noninvasive coronary angiography with multi-slice computed tomography and myocardial perfusion imaging. J Am Coll Cardiol. 2006 Dec 19;48(12):2508-14. doi: 10.1016/j.jacc.2006.05.080. Epub 2006 Nov 28. PMID 17174190
- [Background] Takx RA, Blomberg BA, El Aidi H, Habets J, de Jong PA, Nagel E, Hoffmann U, Leiner T. Diagnostic accuracy of stress myocardial perfusion imaging compared to invasive coronary angiography with fractional flow reserve meta-analysis. Circ Cardiovasc Imaging. 2015 Jan;8(1):e002666. doi: 10.1161/CIRCIMAGING.114.002666. PMID 25596143
- [Background] Yang Z, Zheng H, Zhou T, Yang LF, Hu XF, Peng ZH, Jiang YZ, Li M, Sun G. Diagnostic performance of myocardial perfusion imaging with SPECT, CT and MR compared to fractional flow reserve as reference standard. Int J Cardiol. 2015;190:103-5. doi: 10.1016/j.ijcard.2015.04.091. Epub 2015 Apr 15. No abstract available. PMID 25920018
- [Background] Pontone G, Andreini D, Guaricci AI, Baggiano A, Fazzari F, Guglielmo M, Muscogiuri G, Berzovini CM, Pasquini A, Mushtaq S, Conte E, Calligaris G, De Martini S, Ferrari C, Galli S, Grancini L, Ravagnani P, Teruzzi G, Trabattoni D, Fabbiocchi F, Lualdi A, Montorsi P, Rabbat MG, Bartorelli AL, Pepi M. Incremental Diagnostic Value of Stress Computed Tomography Myocardial Perfusion With Whole-Heart Coverage CT Scanner in Intermediate- to High-Risk Symptomatic Patients Suspected of Coronary Artery Disease. JACC Cardiovasc Imaging. 2019 Feb;12(2):338-349. doi: 10.1016/j.jcmg.2017.10.025. Epub 2018 Feb 14. PMID 29454774
- [Background] Pontone G, Andreini D, Guaricci AI, Guglielmo M, Baggiano A, Muscogiuri G, Fusini L, Soldi M, Fazzari F, Berzovini C, Pasquini A, Ciancarella P, Mushtaq S, Conte E, Calligaris G, De Martini S, Ferrari C, Galli S, Grancini L, Ravagnani P, Teruzzi G, Trabattoni D, Fabbiocchi F, Lualdi A, Montorsi P, Rabbat MG, Bartorelli AL, Pepi M. Quantitative vs. qualitative evaluation of static stress computed tomography perfusion to detect haemodynamically significant coronary artery disease. Eur Heart J Cardiovasc Imaging. 2018 Nov 1;19(11):1244-1252. doi: 10.1093/ehjci/jey111. PMID 30107557
- [Background] Jensen JM, Voss M, Hansen VB, Andersen LK, Johansen PB, Munkholm H, Norgaard BL. Risk stratification of patients suspected of coronary artery disease: comparison of five different models. Atherosclerosis. 2012 Feb;220(2):557-62. doi: 10.1016/j.atherosclerosis.2011.11.027. Epub 2011 Nov 25. PMID 22189201
- [Background] Pontone G, Andreini D, Bertella E, Baggiano A, Mushtaq S, Loguercio M, Segurini C, Conte E, Beltrama V, Annoni A, Formenti A, Petulla M, Guaricci AI, Montorsi P, Trabattoni D, Bartorelli AL, Pepi M. Impact of an intra-cycle motion correction algorithm on overall evaluability and diagnostic accuracy of computed tomography coronary angiography. Eur Radiol. 2016 Jan;26(1):147-56. doi: 10.1007/s00330-015-3793-1. Epub 2015 May 9. PMID 25953001
- [Background] Leipsic J, Abbara S, Achenbach S, Cury R, Earls JP, Mancini GJ, Nieman K, Pontone G, Raff GL. SCCT guidelines for the interpretation and reporting of coronary CT angiography: a report of the Society of Cardiovascular Computed Tomography Guidelines Committee. J Cardiovasc Comput Tomogr. 2014 Sep-Oct;8(5):342-58. doi: 10.1016/j.jcct.2014.07.003. Epub 2014 Jul 24. No abstract available. PMID 25301040
- [Background] Austen WG, Edwards JE, Frye RL, Gensini GG, Gott VL, Griffith LS, McGoon DC, Murphy ML, Roe BB. A reporting system on patients evaluated for coronary artery disease. Report of the Ad Hoc Committee for Grading of Coronary Artery Disease, Council on Cardiovascular Surgery, American Heart Association. Circulation. 1975 Apr;51(4 Suppl):5-40. doi: 10.1161/01.cir.51.4.5. No abstract available. PMID 1116248
- [Background] Andreini D, Pontone G, Bartorelli AL, Trabattoni D, Mushtaq S, Bertella E, Annoni A, Formenti A, Cortinovis S, Montorsi P, Veglia F, Ballerini G, Pepi M. Comparison of feasibility and diagnostic accuracy of 64-slice multidetector computed tomographic coronary angiography versus invasive coronary angiography versus intravascular ultrasound for evaluation of in-stent restenosis. Am J Cardiol. 2009 May 15;103(10):1349-58. doi: 10.1016/j.amjcard.2009.01.343. Epub 2009 Mar 25. PMID 19427427
- [Background] Cury RC, Magalhaes TA, Paladino AT, Shiozaki AA, Perini M, Senra T, Lemos PA, Cury RC, Rochitte CE. Dipyridamole stress and rest transmural myocardial perfusion ratio evaluation by 64 detector-row computed tomography. J Cardiovasc Comput Tomogr. 2011 Nov-Dec;5(6):443-8. doi: 10.1016/j.jcct.2011.10.012. Epub 2011 Nov 4. PMID 22146503
- [Background] Cerci RJ, Arbab-Zadeh A, George RT, Miller JM, Vavere AL, Mehra V, Yoneyama K, Texter J, Foster C, Guo W, Cox C, Brinker J, Di Carli M, Lima JA. Aligning coronary anatomy and myocardial perfusion territories: an algorithm for the CORE320 multicenter study. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):587-95. doi: 10.1161/CIRCIMAGING.111.970608. Epub 2012 Aug 10. PMID 22887690
- [Background] Feuchtner G, Goetti R, Plass A, Wieser M, Scheffel H, Wyss C, Stolzmann P, Donati O, Schnabl J, Falk V, Alkadhi H, Leschka S, Cury RC. Adenosine stress high-pitch 128-slice dual-source myocardial computed tomography perfusion for imaging of reversible myocardial ischemia: comparison with magnetic resonance imaging. Circ Cardiovasc Imaging. 2011 Sep;4(5):540-9. doi: 10.1161/CIRCIMAGING.110.961250. Epub 2011 Aug 23. PMID 21862731
- [Background] Einstein AJ, Moser KW, Thompson RC, Cerqueira MD, Henzlova MJ. Radiation dose to patients from cardiac diagnostic imaging. Circulation. 2007 Sep 11;116(11):1290-305. doi: 10.1161/CIRCULATIONAHA.107.688101. No abstract available. PMID 17846343
- [Background] Moschetti K, Favre D, Pinget C, Pilz G, Petersen SE, Wagner A, Wasserfallen JB, Schwitter JJ. Comparative cost-effectiveness analyses of cardiovascular magnetic resonance and coronary angiography combined with fractional flow reserve for the diagnosis of coronary artery disease. J Cardiovasc Magn Reson. 2014 Jan 25;16(1):13. doi: 10.1186/1532-429X-16-13. PMID 24461028
- [Background] Turchetti G, Lorenzoni V, Bellelli S, Pierotti F, Rovai D, Caselli C, Underwood R, Knuuti J, Neglia D. Effectiveness And Costs Of Different Strategies For The Diagnosis Of Stable Coronary Artery Disease Results From The Evinci Study. Value Health. 2014 Nov;17(7):A474. doi: 10.1016/j.jval.2014.08.1352. Epub 2014 Oct 26. No abstract available. PMID 27201365
- [Background] Hlatky MA, Shilane D, Hachamovitch R, Dicarli MF; SPARC Investigators. Economic outcomes in the Study of Myocardial Perfusion and Coronary Anatomy Imaging Roles in Coronary Artery Disease registry: the SPARC Study. J Am Coll Cardiol. 2014 Mar 18;63(10):1002-8. doi: 10.1016/j.jacc.2013.11.038. PMID 24636556
- [Background] Lubbers M, Coenen A, Kofflard M, Bruning T, Kietselaer B, Galema T, Kock M, Niezen A, Das M, van Gent M, van den Bos EJ, van Woerkens L, Musters P, Kooij S, Nous F, Budde R, Hunink M, Nieman K. Comprehensive Cardiac CT With Myocardial Perfusion Imaging Versus Functional Testing in Suspected Coronary Artery Disease: The Multicenter, Randomized CRESCENT-II Trial. JACC Cardiovasc Imaging. 2018 Nov;11(11):1625-1636. doi: 10.1016/j.jcmg.2017.10.010. Epub 2017 Dec 13. PMID 29248657
- [Background] American College of Cardiology Foundation Task Force on Expert Consensus Documents; Mark DB, Berman DS, Budoff MJ, Carr JJ, Gerber TC, Hecht HS, Hlatky MA, Hodgson JM, Lauer MS, Miller JM, Morin RL, Mukherjee D, Poon M, Rubin GD, Schwartz RS. ACCF/ACR/AHA/NASCI/SAIP/SCAI/SCCT 2010 expert consensus document on coronary computed tomographic angiography: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents. Circulation. 2010 Jun 8;121(22):2509-43. doi: 10.1161/CIR.0b013e3181d4b618. Epub 2010 May 17. No abstract available. PMID 20479158
- [Background] Min JK, Dunning A, Lin FY, Achenbach S, Al-Mallah M, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng V, Chinnaiyan K, Chow BJ, Delago A, Hadamitzky M, Hausleiter J, Kaufmann P, Maffei E, Raff G, Shaw LJ, Villines T, Berman DS; CONFIRM Investigators. Age- and sex-related differences in all-cause mortality risk based on coronary computed tomography angiography findings results from the International Multicenter CONFIRM (Coronary CT Angiography Evaluation for Clinical Outcomes: An International Multicenter Registry) of 23,854 patients without known coronary artery disease. J Am Coll Cardiol. 2011 Aug 16;58(8):849-60. doi: 10.1016/j.jacc.2011.02.074. PMID 21835321
- [Background] Pontone G, Andreini D, Bartorelli AL, Cortinovis S, Mushtaq S, Bertella E, Annoni A, Formenti A, Nobili E, Trabattoni D, Montorsi P, Ballerini G, Agostoni P, Pepi M. Diagnostic accuracy of coronary computed tomography angiography: a comparison between prospective and retrospective electrocardiogram triggering. J Am Coll Cardiol. 2009 Jul 21;54(4):346-55. doi: 10.1016/j.jacc.2009.04.027. PMID 19608033
- [Background] Douglas PS, Hoffmann U. Anatomical versus Functional Testing for Coronary Artery Disease. N Engl J Med. 2015 Jul 2;373(1):91. doi: 10.1056/NEJMc1505594. No abstract available. PMID 26132947
- [Background] Mudrick D, Kaltenbach LA, Shah B, Lytle B, Masoudi FA, Mark DB, Federspiel JJ, Cowper PA, Green C, Douglas PS. Downstream testing and subsequent procedures after coronary computed tomographic angiography following coronary stenting in patients >/=65 years of age. Am J Cardiol. 2012 Sep 15;110(6):776-83. doi: 10.1016/j.amjcard.2012.05.004. Epub 2012 May 30. PMID 22651883
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; ESC Scientific Document Group. Fourth universal definition of myocardial infarction (2018). Eur Heart J. 2019 Jan 14;40(3):237-269. doi: 10.1093/eurheartj/ehy462. No abstract available. PMID 30165617